CLINICAL TRIAL: NCT06570291
Title: A Multicenter, Randomized, Double-blind, Controlled Phase III Trial of Allogenic Adipose Tissue-Derived Mesenchymal Stem Cells (AlloJoin®) Therapy for Knee Osteoarthritis.
Brief Title: Allogenic Adipose-Derived Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuxi Cellular Biopharmaceutical Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBM-MSC-007; NCT05996224 (obsolete NCT alias)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesenchymal stem cells (Experimental)
  Interventions: Drug: Mesenchymal Stem Cells
- Sodium hyaluronate (Placebo Comparator)
  Interventions: Drug: Sodium Hyaluronate Injection

INTERVENTIONS:
Drug: Mesenchymal Stem Cells — Allogenic adipose tissue-derived mesenchymal stem cells administrated for intra- articular use
  Arms: Mesenchymal stem cells
Drug: Sodium Hyaluronate Injection — Sodium Hyaluronate administrated for intra-articular use
  Arms: Sodium hyaluronate

SUMMARY:
Evaluate the efficacy and safety of Allogenic Adipose Tissue-Derived Mesenchymal Stem Cells Therapy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and voluntarily sign the consent form before this study；
2. According to the diagnostic criteria (American Rheumatology Association, clinical + radiology criteria), patients with knee osteoarthritis are definitely diagnosed；Course of knee osteoarthritis was more than 6 months;
3. Age: 40-75, males and females；
4. The subjects' WOMAC score was 24-72
5. The Kellgren Lawrence grade (X-ray axial position of knee joint) of subjects was grade II / III;
6. Subjects are generally in good condition and can walk autonomously, except for those who use wheelchairs, walking aids or crutches.

Exclusion Criteria:

1. The subject may be allergic to the main cell preparation components (B vitamins, amino acids and so on).
2. The subject received systemic and / or local treatment with autologous and / or allogeneic mesenchymal progenitor cells.
3. The subject considered obese.
4. Laboratory test (any item meets): neutrophil absolute number < 1.0 × 10^9 / L, platelet count < 50 × 10^9 / L, serum albumin < 30g / L, serum creatinine > upper limit of 1.2 times normal value range, total bilirubin、alanine aminotransferase、aspartate aminotransferase > upper limit of 2 times of normal value range.
5. The subject has diseases or symptoms may affect VAS, WOMAC and so on.
6. The subject has serious and poorly controlled concomitant diseases, such as (but not limited to) nervous system, cardiovascular, liver, kidney, gastrointestinal and endocrine diseases, which may prevent the subjects from participating in the study according to the judgment of the researchers.
7. The subject has an history malignant tumour.
8. The subject has connective tissue disease or rheumatoid arthritis、chondropathy、Chondrocalcinosis articularis、 Hemochromatosis、inflammatory arthropathy、avascular necrosis of femoral head、Paget's disease、hemophilic arthropathy、infectional arthritis、Charcot' s disease、villonodular synovitis or synovial chondromatosis.
9. The subject has severe generalized infectious diseases or local knee infection (including skin and intra-articular infection) in the 3 months prior to this trial.
10. According to the researchers, the subject has disease of lower limbs which may be interfered knee evaluation, for example fibromyalgia, osphyalgia, lumbar disc protrusion and so on.
11. The subject had any other coagulation dysfunction caused by acute or chronic diseases, according to the judgment of the researchers, this coagulation dysfunction may endanger the safety of patients and / or affect the judgment of knee joint evaluation indicators.
12. The subject has received arthroscopic surgery or other open surgery related to knee joint operation in the 6 months prior to this trial.
13. The subject has received other intra-articular injections, including but not limited to hyaluronic acid, hormone, PRP, BMP (bone morphogenetic protein) , hypertonic glucose and so on for KOA in the 3 months preceding the trial.
14. The subject has received aminoglucose or chondroitin sulfate within 1 month before the treatment.
15. The subject has used dexamethasone, prednisone, hydrocortisone and other hormones orally / intravenously within 1 month before the treatment.
16. The subject has attenuated or live attenuated vaccine injection with 1 month before the treatment.
17. The subject has undergone knee prosthesis or a plan of knee prosthesis within the trial.
18. The subject has contraindication of MRI, included but not only: the subject installed heart pacemaker, defibrillator, heart bracket, heart valve prosthesis, metal clip after aneurysm surgery, drug infusion device implanted in vivo, any electronic device implanted in the body (nerve stimulator, bone growth stimulator) endovascular coil, strainer, ECG monitor, metal suture, shrapnel or sand of body, plate fixation and steel nail after fracture surgery, artificial cochlea, middle ear shift plant, metallic intraocular foreign body etc; the subject is a claustrophobia, critical ill patient and so on.
19. The subject tests positive for: HIV, HBV, HCV and treponema pallidum.
20. The subject has history of alcoholism, drug abuse, or mental illness in the 3 years prior to this trial.
21. The subject has participated in any other clinical trial in the 3 months prior to this trial.
22. The subject (including male subjects) has fertility, sperm donation or egg donation plans during the trial period; the female subject is pregnant, lactating or having a positive pregnancy test.
23. The subject is legally disabled by reference to the law of the people's Republic of China on the protection of disabled persons (April 2008).
24. The subject has any other unsuitable condition (such as factors reducing the follow-up compliance) to be determined by the investigator.
25. The Kellgren Lawrence grade (X-ray axial position of knee joint) of any knee joint of the subjects was grade IV.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC score | 48 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index;0-96 points；96 points mean a worse outcome,will be tested at 48 weeks after the first injection
MRI quantitative analysis of articular cartilage | 24 weeks

SECONDARY OUTCOMES:
WOMAC Score | 4、12、24、36、60、72、84 and 104 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index;0-96 points；96 points mean a worse outcome, will be tested at 4、12、24、36、60、72、84 and 104 weeks after the first injection
MRI quantitative analysis of articular cartilage （volume change percentage） | 12、48、104 weeks
  Magnetic Resonance Imaging analysis of articular cartilage, will be tested at 12、48、104 weeks after the first injection
MRI quantitative analysis of articular cartilage (volume change) | 12、24、 48 and 104 weeks
  Magnetic Resonance Imaging analysis of articular cartilage, will be tested at 12、24、 48 and 104 weeks after the first injection
VAS Score | 4、12、24、36、48、60、72、84、104 weeks
  Visual Analogue Scale/Score；0-10 points；10 points mean the worse outcome,will be tested at 4、12、24、36、48、60、72、84 and 104 weeks after the first injection
SF-36 | 4、12、24、36、48、60、72、84、104 weeks
  The Medical Outcomes Study 36-Item Short-Form Health Survey;0-100 points；100 points mean a better outcome, will be tested at 4、12、24、36、48、60、72、84 and 104 weeks after the first injection
Whole-Organ Magnetic Resonance Imaging Score | 12、24、48 and 104 weeks
  Whole-Organ Magnetic Resonance Imaging Score(WORMS) of the knee; 0-332points; 332 points means the worst outcome; will be assessed at 12、24、48 and104 weeks
mJSW | 104 weeks
  Minimum joint space width (mJSW) of the knee, will be measured at baseline and 104 weeks
Physical examination | Day 0、week 1、2、3、4、12、24、36、48、60、72、84、104 weeks
  Height and weight will be tested and combined to report BMI in kg/m^2at Day 0 and week 1、2、3、4、12、24、36、48、60、72、84、104 weeks
Adverse Events and Serious Adverse Events | Day 0 to 104 weeks
  AE and SAE, will be assessed within the 104 week time span

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - RenJi Hospital, Shanghai, China
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No